CLINICAL TRIAL: NCT05703113
Title: The Effect of the Education Given to Nursing Students With Web 2.0 Tools on the Level of Participation, Attitude, Interest and Motivation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, Metin Yildiz, Nurse (Asst.Prof.Dr.), Sakarya University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SakaryaU-metinyildiz-003
Record Dates: First submitted 2023-01-16; First posted 2023-01-27 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Educational Problems
Keywords: Web 2.0 tools; participation; attitude; interest; motivation
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group trained with Web 2.0 tools (Experimental): Group trained with Web 2.0 tools: Web 2.0 tools were used both while making presentations to the students and at the time of evaluation. Wordaart, google form, padlet, canva, bubbl.us were used in the presentation as Web 2.0 tools. For reviews kahoot, Socrative, Bamboozle, Mentimeter and Who Wants To Be A Millionaire? application is used.
  Interventions: Behavioral: Web 2.0 tools
- Control Group (No Intervention): Lessons were taught with traditional learning method.

INTERVENTIONS:
Behavioral: Web 2.0 tools — Education with Web 2.0 tools
  Arms: Group trained with Web 2.0 tools

SUMMARY:
In this study, it is aimed to examine the effects of the education given to nursing students with web 2.0 tools on students' participation, attitude, interest and motivation levels.

The research was conducted as a randomized controlled experimental study. The study population consisted of 150 students between October 2022 and January 2023, and the sample of the research consisted of 110 individuals selected from the population using the improbable random sampling method. "Descriptive Feature Form," "Teaching Material Motivation Scale," "Course Interest Scale", Attitude Scale Towards Learning and ''absence charts'' were used to collect data.

In the analysis of data; percentile distribution, chi-square, Fisher- Exact test, t-test in independent groups, paired samples t Test were used.

ELIGIBILITY:
Inclusion Criteria:

* To be a student,
* 18 years and older
* Volunteer

Exclusion Criteria:

* Students who are not required to attend the course are not included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-01-15 (Actual)

PRIMARY OUTCOMES:
Teaching Material Motivation Scale | Evaluated at the end of 6 weeks.
  Teaching Material Motivation Scale Teaching Material Motivation Instructional Material Motivation Scale: It was developed to measure the effect of instructional materials on students' motivation. The scale is a 5-point Likert-type scale consisting of 36 items. Each item in the scale will be scored from 1 (Not True) to 5 (Very True) by the students. Accordingly, the lowest score on the scale is 36, and the highest score is 180. An increase in the score on the scale indicates an increase in motivation.
Student Interest Scale | Evaluated at the end of 6 weeks.
  Student Interest Scale:
  Student Interest Scale; Developed by (Mazer, 2013) in order to evaluate its relationship with variables such as learning motivation, effective learning, and level of participation in the lesson, the Class Interest Scale is a 5-point Likert-type measurement tool consisting of 16 items and two sub-dimensions (affective and cognitive interest). et al (2015) ("1" Strongly disagree, "2" Disagree, "3" Undecided, "4" Agree, "5" Totally Agree). There is no reverse coded item in the scale. Affective interest sub-dimension of the scale consists of 9 items and cognitive interest sub-dimension consists of 7 items. As the scale score increases, the interest increases.
Attitude Scale Towards Learning | Evaluated at the end of 6 weeks.
  Attitude Scale Towards Learning:Attitude Scale Towards Learning: The scale developed by Çetin et al. was developed to determine students' attitudes. As a result of all validity and reliability analyzes, there are 34 items in total. Of these scale items, 25 are positive and 9 are negative. The five-point Likert scale is "Totally Agree", "Strongly Agree", "Partly Agree", "Disagree", "Strongly Disagree". The highest attitude score that can be obtained from the scale is 170 and the lowest attitude score is 34. As the attitude score increases, the positive attitude increases.
Class participation | Evaluated at the end of 6 weeks.
  Class participation:A weekly signature chart was taken from the students and the number of absenteeism in the last week was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Metin YILDIZ, Asst.Prof.Dr., Principal Investigator — Sakarya University
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)